CLINICAL TRIAL: NCT00147784
Title: HEPMET-1: Evaluate the Feasibility, Mental Sideeffects and the Efficacy of Hepatitis C Treatment in a Methadone Maintenance Treated (MMT) Opioid Addicted Group.
Brief Title: HEPMET-1: Evaluate the Feasibility, Mental Sideeffects and the Efficacy of Hepatitis C Treatment in a MMT Group.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Oistein Kristensen, MD, Sorlandet Hospital HF
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSHF-70332; Protocol no 9772387; EudraCT no 2005-002869-37
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Opiate Dependence; Hepatitis
Keywords: Chronical Hepatitis C treatment; Methadone Maintenance Treatment; Pegylated Interferon and Ribavirin; 14 weeks treatment; Genotype 2 and 3
MeSH Terms: conditions — Opioid-Related Disorders; Hepatitis | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin — 800 mg pr. os daily, 400 mg morning and 400 mg evening (200 mg/tbl.) for 14 weeks
Drug: Pegylated Interferon — 180 mikrogram in 0,5 ml solution s.c. once a week for 14 weeks

SUMMARY:
* To evaluate if weekly psychological follow-up make opioid dependent patients in MMT able to accomplish 14 weeks treatment with Peginterferon alfa-2a (PEG-INF) and ribavirin to the same extent than non-opioid dependents.
* To determine the efficacy of this anti-HCV treatment

DETAILED DESCRIPTION:
Chronic infection with the hepatitis C virus (HCV) is a health problem worldwide. In Norway, there are about 3000 patients participating in Methadone Maintenance Treatment(MMT) programs. A prevalence study at the MMT treatment unit in Kristiansand, showed that more than 90 % of 177 patients have been infected with hepatitis C.

A major problem with anti-HCV treatment for this group is the lack of compliance and retention in treatment. Further, due to the high incidence of psychological disorders in opioid dependent patients, this may also complicate anti-HCV treatment. Drug addicted in MMT treatments programs may find themselves excluded from Hepatitis C treatment.

Due to better treatment efficacy with the new PEG-INF's and encouraging reports from 14 weeks studies, it may be easier to motivate opioid dependents to fulfill treatment. Weekly psychological follow-up of these patients will further increase the possibility of opioid dependents in MMT to be able to complete anti-HCV treatment.

The aim of this study is to focus on this patients situation, and strengthen their possibility to have a real opportunity to get treatment. We therefore wish to make a pilot study to investigate the feasibility, efficacy and psycological side-effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of hepatitis C infection, genotype 2 and 3
* Normal or elevated serum ALT activity
* In MMT-programme and with at least 6 months with satisfactory drug abuse control. That means no iv injections and no or minimal use of drugs.
* Male and female patients

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Untreated serious psychiatric disorders, particularly depression.
* Serious drug abuse or alcohol abuse last 6 months
* Intravenous drug abuse last 6 months
* Hepatitis A, B or HIV infection
* HCV genotype 1, 4, 5 and 6
* Leucocytes < 3000 cells/mm3 at screening (neutrophil count <1500 cells/mm3)
* Platelet count < 80 000 cells/mm3 at screening
* Hb <11 g/dL in women or <12 g/dL in men at screening
* Documented or presumed coronary artery disease or cerebrovascular disease
* Thyroid dysfunction not adequately controlled
* Epilepsy
* Malignant disease

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
- Percent of patients with sustained virological response, defined as undetectable HCV RNA 24 weeks after end of treatment | 24 weeks after end of treatment

SECONDARY OUTCOMES:
Retention in treatment, compliance, psychological distress, measures of quality of life, perceived drug use control and urine toxicology | 2, 4, 8, 14 and 24 weeks after study start

CONTACTS AND LOCATIONS:
Overall Officials: Oistein Kristensen, MD, Principal Investigator — Soerlandet Hospital HF; Oistein Kristensen, MD, Principal Investigator — Addiction Unit, SSHF
Locations (2):
- Norway (2):
  - Soerlandet Hospital HF, Kristiansand, Vest-Agder
  - Addiction Unit, Sorlandet Hospital, Kristiansand, Vest-Agder

REFERENCES:
- [Derived] Kristensen O, Sundoy A, Skeie K, Vederhus JK, Oye I, Opsal A, Rysstad O, Gallefoss F. [Short-term treatment of Hepatitis C in heroin-dependent patients]. Tidsskr Nor Laegeforen. 2009 Aug 27;129(16):1639-42. doi: 10.4045/tidsskr.09.33690. Norwegian. PMID 19721480